CLINICAL TRIAL: NCT06471881
Title: Clinical and Radiographical Performance of Zirconia Bars for Mandibular Implant Overdentures: A 3-year Follow-up Prospective Cohort Study
Brief Title: Zirconia Bars for Mandibular Implant Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zirconia bars
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Edentulous Mouth
Keywords: Cohort study; Edentulism; Implant overdentures; Zirconia; Prosthodontic maintenance; Dental implants
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zirconia bars with distal extensions (Experimental): Two mandibular implants and a mandibular implant overdenture supported by a computer-aided design
  Interventions: Device: Two mandibular implants

INTERVENTIONS:
Device: Two mandibular implants — Rehabilitation with two mandibular implants and a mandibular implant overdenture supported by a computer-aided design bar

SUMMARY:
Purpose: To assess the clinical and radiographic outcomes of computer-aided designed and manufactured (CAD-CAM) zirconia bars supporting mandibular implant-retained overdentures (IODs) after a 3-year follow-up.

Methods: A prospective observational single-center study involving 30 edentulous patients rehabilitated with two mandibular implants and a mandibular implant overdenture supported by a computer-aided design - computer-assisted manufacturing zirconia bar with distal extensions was performed assessing clinical and radiographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous individuals for more than one year.
* Individuals with sufficient anatomical bone conditions in the interforaminal area to place implants of 4.3mm in diameter and at least 10.0mm in length without bone augmentation needs.
* Written consent to participate and to attend the study and the yearly follow-ups.

Exclusion Criteria:

* Individuals suffered from psychiatric problems.
* History of cerebrovascular or cardiovascular accident within the last six months.
* Uncontrolled or insulin-dependent diabetes, immuno-compromised status, current chemotherapy, and leukocyte system diseases.
* Severe systemic health conditions do not allow surgical intervention with local anesthesia.
* Irradiated bone.
* Severe parafunctional habits
* Drugs or alcohol abuse.
* Insufficient oral hygiene.
* Unrealistic treatment demands.
* Smokers were not excluded, but a cessation protocol was suggested before the implant treatment.
* Unwillingness to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Implant Survival | 36 months
  Number of patients with continued presence of the implant(s) during the re-examination appointments
Implant Success | 36 months
  Number of patients with absence of persisting subjective discomfort such as pain, foreign body perception and or dysesthesia (i.e., painful sensation), absence of a recurrent peri-implant infection with suppuration, absence of implant mobility on manual palpation, absence of any continuous peri-implant radiolucency
Prosthetic Survival | 36 months
  Number of patients with functional presence of the denture and the bar at the follow-up moments
Prosthetic Success | 36 months
  Number of patients with absence of any technical/mechanical complications without the need to repair the dentures (including the attachment systems) or the bars
Radiological evaluation | 36 months
  Marginal bone loss
Radiological examination | 36 months
  Implant bar fit

CONTACTS AND LOCATIONS:
Overall Officials: Joannis Katsoulis, Prof., Study Director — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molinero-Mourelle P, Fonseca M, Grossen ME, Zuercher AN, Schimmel M, Katsoulis J. Clinical and Radiographic Evaluation of Zirconia Bars for Mandibular Implant Overdentures: A Prospective Cohort Study With up to 3 Years of Follow-Up. Clin Implant Dent Relat Res. 2025 Aug;27(4):e70066. doi: 10.1111/cid.70066. PMID 40709726